CLINICAL TRIAL: NCT04342702
Title: A Study on the Prospective Cohort Library of Novel Coronavirus Pneumonia in Southeran
Brief Title: A Study on the Prospective Cohort Library of COVID-19 in Southeran
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Wenzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Wenzhou Central Hospital And Sixth People's Hospital of Wenzhou Medical University (Unknown); Yueqing Hospital of Wenzhou Medical University (Unknown); Ruian Hospital of Wenzhou Medical University (Unknown); Cangnan Hospital of Wenzhou Medical University (Unknown); Pingyang Hospital of Wenzhou Medical University (Unknown); Yongjia People's Hospital (Unknown)
Responsible Party: Principal Investigator, Xiaokun Li, Professor, Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2020-NCP-202
Record Dates: First submitted 2020-04-04; First posted 2020-04-13 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Follow-up; COVID-19; Infectious Diseases; Respiratory
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre population-based follow-up study for all 504 patients with laboratory-confirmed COVID-19. This study establishes a standardized and structured clinical database to provide complete and multidimensional clinical diagnosis and treatment data of novel coronavirus pneumonia, which also support future epidemiological, infectious disease study and patients' prognosis, by collecting clinical data and the related data of patients with novel coronavirus pneumonia in Southern Zhejiang province.

DETAILED DESCRIPTION:
The follow-up information will be collected in one-month, three-month, six-month and one-year after discharge. Information about symptoms, radiographic and laboratory findings, lung function, SF-36 QUESTIONNAIRE, antibody of COVID19，result of RT-PCR Test and suvival information will be collected through all time frames.

ELIGIBILITY:
Inclusion Criteria:

* All patients with laboratory-confirmed COVID-19 in Wenzhou

Exclusion Criteria:

* Suspected cases of COVID-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Among all 504 patients with laboratory-confirmed COVID-19, 190 patients were classified as the imported cohort, and 311 patients were classified into the secondary cohort, three patients were excluded. The patients' inclusion cutoff was March 15, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
36-Item Short Form Survey Instrument (SF-36) | one month, three month, six month and one year after discharge, minimum score
  sum score of SF 36 form in each time frame
the value of FEV1 by lung function test | one month, three month, six month and one year after discharge
the ratio of FEV1 to FVC by lung function test | one month, three month, six month and one year after discharge

SECONDARY OUTCOMES:
the predicted value of FEV1 by lung function test | one month, three month, six month and one year after discharge
the predicted ratio of FEV1 to FVC by lung function test | one month, three month, six month and one year after discharge
Lymphocyte value | one month, three month, six month and one year after discharge
  laboratory result
Neutrophil value | one month, three month, six month and one year after discharge
  laboratory result
DDI value | one month, three month, six month and one year after discharge
  laboratory result
the proportion of applying ACEIs/ARBs medication | from the date of hospital admission to the day of hospital discharge
  collect the number of applying ACEIs/ARBs medication and calculate the proportion
number of clinical symptoms after hospital discharge | one month, three month, six month and one year after discharge
  clinical symptoms
number of cases returning to positive result in RT-PCR test | one month, three month, six month and one year after discharge
Number of positive outcome of IgG for antibody of COVID-19 | one month, three month, six month and one year after discharge

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang